CLINICAL TRIAL: NCT01865448
Title: Study to Assess the Effects of DHA (Docosahexaenoic Acid) on Pro-resolving Anti-inflammatory Mediators in Obese Patients Undergoing Weight-loss Treatment
Brief Title: Effects of DHA on Pro-resolving Anti-inflammatory Mediators in Obese Patients Undergoing Weight-loss Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Protein Supplies SL (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PNK-DHA-2013-01
Record Dates: First submitted 2013-05-27; First posted 2013-05-30 (Estimated); Results first posted 2019-06-20 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-03

CONDITIONS: Obesity; Inflammation
Keywords: Docosahexaenoic Acids; Fatty Acids, Omega-3; Obesity; Inflammation
MeSH Terms: conditions — Obesity; Inflammation | interventions — Docosahexaenoic Acids; Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- omega-3 DHA (Active Comparator): Patients in this group will receive 500 mg/day supplement of DHA omega-3 fatty acid in capsule form, in addition to the vitamin and oligoelement supplements which are part of the standard weight-loss programme.
  Interventions: Dietary Supplement: Omega-3 DHA
- Control (Placebo Comparator): Patients in control group will receive an placebo capsule, in addition to the vitamin and oligoelement supplements which are part of the standard weight-loss programme
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Omega-3 DHA — Patients take daily 2 tablets of Docosahexaenoic Acid
  Other Names: Docosahexaenoic Acid; omega-3 fatty acid; PUFA
  Arms: omega-3 DHA
Other: Placebo — Patients in control group take daily 2 placebo capsule
  Other Names: placebo capsule
  Arms: Control

SUMMARY:
Comparative, randomized, placebo-controlled, single-centre, single-blind clinical trial to assess the effectiveness of providing additional DHA omega-3 fatty acids supplements to increase the levels of pro-resolving and anti-inflammatory lipid mediators and decrease the biological markers of chronic inflammation in obese patients following a weight-loss programme.

DETAILED DESCRIPTION:
Will include obese patients (BMI between 30 and 35) who are following a standardized, multidisciplinary weight-loss programme (PronoKal® Method), which consists of a very-low-calorie diet based on protein packets and vegetables with a low glycemic index, into which natural foods are gradually reintroduced, accompanied by physical exercise and emotional support.

Patients who are being treated with acetylsalicylic acid (ASA), non-steroidal anti-inflammatory drugs (NSAIDS), corticoids or thiazolidinedione antidiabetic drugs (glitazones); and patients with immune disorders (rheumatoid arthritis, Lupus, etc.) and/or inflammatory disease (ulcerative colitis, Crohn's disease, etc.) who may alter the biological markers of inflammation,will be excluded.

Treatment: In addition to the vitamin and oligoelement supplements which are part of the standard weight-loss programme, the patients will receive an additional 500 mg/day supplement of DHA omega-3 fatty acids in capsule form (study group) or a placebo capsule (control group).

The follow up will be 6 months and patients will be monitored over the course of 6 control visits: baseline, 7 days, 15 days, 30 days, 60 days and 180 days.

The main objective is to assess the effectiveness of providing additional DHA supplements to increase the levels of pro-resolving and anti-inflammatory lipid mediators and decrease the biological markers of chronic inflammation in obese patients following a weight-loss programme.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* Obese patients with Body Mass Index between 30 and 35
* Patients who, regardless of their inclusion in this study, are going to follow the standardized weight-loss programme (PronoKal® Method)
* Patients who agree to participate and sign the Informed Consent form

Exclusion Criteria:

* Treatment with Omega-3 fatty acid supplements for other reasons during the month prior to inclusion in the trial
* Treatment with acetylsalicylic acid (ASA), non-steroidal anti-inflammatory drugs (NSAIDS), corticoids or thiazolidinedione antidiabetic drugs (glitazones)
* Pregnant or nursing patients
* Haemopathy, including clotting disorders
* Treatment with dicoumarin anticoagulants (Sintrom®)
* Cancer or a history of cancer who have not received the oncologist's release
* Type 1 or type 2 diabetes mellitus
* Immune disorders (rheumatoid arthritis, lupus, etc.) and/or inflammatory disease (ulcerative colitis, Crohn's disease, etc.) that may alter the biological markers of inflammation
* Patients not expected to attend monitoring visits

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-05; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel De Luis, PhD, Principal Investigator — Unidad de Apoyo a la Investigacion. Hospital Rio Hortega
Locations (1):
- Research Support Unit. Río Hortega University Hospital, Valladolid, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study performed in a single center. The patients attending the Endocrinology and Nutrition Department at the Hospital Clinico Universitario of Valladolid to receive treatment for obesity were consecutively enrolled in this study.
Groups:
- Control: Patients in this group will receive an placebo capsule, in addition to the vitamin and oligoelement supplements which are part of the standard weight-loss programme
- Omega-3 DHA: Patients in this group will receive 500 mg/day supplement of DHA omega-3 fatty acid in capsule form, in addition to the vitamin and oligoelement supplements which are part of the standard weight-loss programme.
  Omega-3 DHA: Patients take daily 2 tablets of placebo
Period: Overall Study
Arm/Group | Control | Omega-3 DHA
Started | 17 | 17
Completed | 15 | 14
Not Completed | 2 | 3
Not completed — Adverse Event | 1 | 1
Not completed — Pregnancy | 0 | 1
Not completed — dropout unrelated to study | 1 | 1

BASELINE CHARACTERISTICS:
Population: Analysis with completers only
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Omega-3 DHA | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (11.7) | 47.4 (9.1) | 45.8 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 7 | 5 | 12
Region of Enrollment [Number; unit: participants]
  Spain | 15 | 14 | 29
Weight (Kg) [Mean (Standard Deviation); unit: Kg] | 92.2 (13.1) | 92.1 (8.7) | 92.1 (10.9)
Body Mass Index (BMI) (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 32.9 (1.9) | 33.4 (1.4) | 33.1 (1.6)
Waist circumference (cm) [Mean (Standard Deviation); unit: cm] | 109.2 (7.9) | 109.4 (7.8) | 109.3 (7.7)
15-HETE [Mean (Standard Deviation); unit: pg/ml] | 51.14 (84.24) | 23.76 (38.35) | 36.9 (64.8)
12 -HETE [Mean (Standard Deviation); unit: pg/ml] | 4985.94 (4301.86) | 5359.26 (3431.47) | 5179.51 (3803.27)
8-HETE [Mean (Standard Deviation); unit: pg/ml] | 43.74 (42.24) | 57.85 (51.38) | 51.06 (46.85)
5-HETE [Mean (Standard Deviation); unit: pg/ml] | 424.39 (209.93) | 369.63 (106.82) | 396.00 (163.78)
TXB2 [Mean (Standard Deviation); unit: pg/ml] | 118.20 (133.33) | 131.26 (95.62) | 124.97 (113.2)
PGE2 [Mean (Standard Deviation); unit: pg/ml] | 2.82 (6.93) | 0.14 (0.34) | 1.43 (4.91)
LTB4 [Mean (Standard Deviation); unit: pg/ml] | 15.08 (29.88) | 0.00 (0.00) | 7.26 (21.71)
17-HDOHE [Mean (Standard Deviation); unit: pg/ml] | 96.56 (87.70) | 133.92 (80.78) | 115.93 (84.70)
14-HDOHE [Mean (Standard Deviation); unit: pg/ml] | 3668.74 (3540.69) | 4071.54 (3150.66) | 3877.60 (3285.03)
7-HDOHE [Mean (Standard Deviation); unit: pg/ml] | 128.55 (52.83) | 120.83 (49.09) | 124.55 (50.08)
4-HDOHE [Mean (Standard Deviation); unit: pg/ml] | 268.36 (148.25) | 288.93 (147.32) | 279.03 (145.27)
RVD2 [Mean (Standard Deviation); unit: pg/ml] | 64.89 (74.55) | 50.68 (91.41) | 57.52 (82.44)
PD1 [Mean (Standard Deviation); unit: pg/ml] | 6.27 (7.04) | 3.80 (5.27) | 4.99 (6.19)
Sum of proinflammatory mediators [Mean (Standard Deviation); unit: pg/ml] — Sum of metabolite mediators derived from arachidonic acid (AA)
  pg/ml | 5641.30 (4357.98) | 5941.89 (3563.60) | 5797.16 (3890.83)
Sum of proresolving mediators [Mean (Standard Deviation); unit: pg/ml] — Sum of PUFA metabolite mediators derived from docosahexaenoic acid (DHA)
  pg/ml | 4233.38 (3652.42) | 4669.69 (3334.98) | 4459.61 (3430.36)
Proresolution index [Mean (Standard Deviation); unit: ratio] — Ratio of summation of proresolving mediators to summation of proinflammatory mediators
  ratio | 0.72 (0.23) | 0.78 (0.35) | 0.75 (0.29)
C-reactive Protein (CRP) (mg/dl) [Mean (Standard Deviation); unit: mg/dl] | 3.3 (1.4) | 3.8 (3.4) | 3.6 (2.5)
Adiponectin (ng/ml) [Mean (Standard Deviation); unit: ng/ml] | 8.6 (4.2) | 7.9 (3.5) | 8.3 (3.8)
Resistin (ng/ml) [Mean (Standard Deviation); unit: ng/ml] | 5.3 (3.6) | 4.5 (2.2) | 4.9 (2.9)
Tnf alpha (ng/ml) [Mean (Standard Deviation); unit: ng/ml] | 4.7 (2.3) | 5.0 (2.5) | 4.8 (2.3)
Interleukin-6 (ng/ml) [Mean (Standard Deviation); unit: ng/ml] | 4.2 (2.1) | 4.1 (1.7) | 4.2 (1.8)
Leptin (ng/ml) [Mean (Standard Deviation); unit: ng/ml] | 29.7 (17.7) | 45.2 (22.4) | 37.2 (21.2)
7SMAR1 [Mean (Standard Deviation); unit: pg/ml] — Baseline 7SMAR1 was below limits of detection
  pg/ml | NA (NA) — Baseline 7SMAR1 was below limits of detection | NA (NA) — Baseline 7SMAR1 was below limits of detection | NA (NA) — Baseline 7SMAR1 was below limits of detection
7RMAR1 [Mean (Standard Deviation); unit: pg/ml] — Baseline 7RMAR1 was below limits of detection
  pg/ml | NA (NA) — Baseline 7RMAR1 was below limits of detection | NA (NA) — Baseline 7RMAR1 was below limits of detection | NA (NA) — Baseline 7RMAR1 was below limits of detection

OUTCOME MEASURES:

1. Primary Outcome: Proresolution Index
Description: Proresolution index is the ratio of sum of proresolving mediators/sum of proinflammatory mediators
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
ratio | 0.71 (0.27) | 0.84 (0.36)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.2780, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p = 0.8689, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p = 0.4533, Paired t-test

2. Secondary Outcome: Weight at 6 Months
Description: Weight at 6 months (end of the monitoring period)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
kg | 71.8 (11.4) | 72.3 (7.1)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.71833, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p < 0.001, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Body Mass Index at 6 Months
Description: Body mass index at 6 months (end of the monitoring period)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
kg/m^2 | 25.6 (1.8) | 26.2 (1.6)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.51900, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p < 0.001, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p < 0.001, Paired t-test

4. Secondary Outcome: Waist Circumference at 6 Months
Description: Waist circumference at 6 Months (end of the monitoring period)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
cm | 87.3 (7.4) | 89.0 (5.2)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.24567, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p < 0.001, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p < 0.001, Paired t-test

5. Primary Outcome: Sum of Proresolving Mediators at 6 Months
Description: Sum of proresolving mediators at 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
pg/ml | 3342.11 (4132.21) | 3409.31 (2065.58)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.9573, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p = 0.5257, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p = 0.0657, Paired t-test

6. Primary Outcome: Sum of Proinflammatory Mediators at 6 Months
Description: Sum of proinflammatory mediators at 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
pg/ml | 4276.89 (35.89) | 3931.00 (1654.83)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.7474, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p = 0.3745, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p = 0.0476, Paired t-test

7. Secondary Outcome: C-reactive Protein (CRP) at 2 Months
Description: Level of c-reactive protein (CRP) at 2 months
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
mg/dl | 2.3 (2.3) | 3.2 (2.9)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.27444, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p < 0.001, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p < 0.001, Paired t-test

8. Secondary Outcome: C-reactive Protein (CRP) at 6 Months
Description: Level of c.reactive protein (CRP) at 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
mg/dl | 1.9 (1.4) | 2.1 (1.2)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.28489, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p < 0.001, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Test type: Superiority or Other; p < 0.001, Paired t-test

9. Secondary Outcome: Adiponectin at 2 Months
Description: Level of Adiponectin at 2 months
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
ng/ml | 11.3 (4.9) | 8.6 (2.6)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.04491, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p < 0.001, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p < 0.001, Paired t-test

10. Secondary Outcome: Adiponectin at 6 Months
Description: Level of Adiponectin at 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
ng/ml | 9.9 (4.8) | 7.9 (3.4)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.24396, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p = 0.00162, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p = 0.00162, Paired t-test

11. Secondary Outcome: Tnf Alpha at 2 Months
Description: Level of Tnf alpha at 2 months
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
ng/ml | 3.1 (2.1) | 3.3 (1.8)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.82322, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p = 0.25908, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p = 0.25908, Paired t-test

12. Secondary Outcome: Tnf Alpha at 6 Months
Description: Level of Tnf alpha at 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
ng/ml | 2.0 (0.4) | 2.0 (0.3)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.76435, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p = 0.18876, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p = 0.18876, Paired t-test

13. Secondary Outcome: Interleukin-6 at 2 Months
Description: Level of Interleukin-6 at 2 months
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
ng/ml | 4.0 (2.1) | 4.3 (1.5)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.40485, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p < 0.001, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p < 0.001, Paired t-test

14. Secondary Outcome: Interleukin-6 at 6 Months
Description: Level of Interleukin-6 at 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
ng/ml | 6.3 (2.7) | 4.9 (2.0)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.13911, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p = 0.05726, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p = 0.05726, Paired t-test

15. Secondary Outcome: Resistin at 2 Months
Description: Level of Resistin at 2 months
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
ng/ml | 4.7 (2.5) | 4.5 (1.9)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.60214, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p < 0.001, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p < 0.001, Paired t-test

16. Secondary Outcome: Resistin at 6 Months
Description: Level of Resistin at 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
ng/ml | 3.6 (2.4) | 3.4 (1.6)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.66053, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p < 0.001, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p < 0.05, Paired t-test

17. Secondary Outcome: Leptin at 2 Months
Description: Level of Leptin at 2 months
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
ng/ml | 5.8 (6.0) | 8.5 (7.1)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.28743, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p < 0.001, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p < 0.001, Paired t-test

18. Secondary Outcome: Leptin at 6 Months
Description: Level of Leptin at 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
ng/ml | 10.2 (5.7) | 15.8 (10.2)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.58561, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p < 0.001, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Test type: Superiority or Other; p < 0.001, Paired t-test

19. Secondary Outcome: 15-HETE at 2 Months
Description: Level of 15-HETE at 2 months
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
pg/ml | 101.37 (136.54) | 49.51 (49.77)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.1953, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p = 0.0351, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p = 0.0795, Paired t-test

20. Secondary Outcome: 15-HETE at 6 Months
Description: Level of 15-HETE at 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
pg/ml | 65.65 (32.65) | 72.95 (51.50)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.6664, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p = 0.4310, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p = 0.0049, Paired t-test

21. Secondary Outcome: 12-HETE at 2 Months
Description: Level 12-HETE at 2 months
Time Frame: 2 month
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
pg/ml | 6526.37 (3922.55) | 5148.86 (1817.86)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.2470, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p = 0.2755, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p = 0.8226, Paired t-test

22. Secondary Outcome: 12-HETE at 6 Months
Description: Level of 12-HETE at 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
pg/ml | 3652.28 (3488.85) | 3226.87 (1431.22)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.6779, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p = 0.3761, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p = 0.0281, Paired t-test

23. Secondary Outcome: 8-HETE at 2 Months
Description: Level of 8-HETE at 2 months
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- Control: Patients in this group will receive an placebo capsule, in addition to the vitamin and oligoelement supplements which are part of the standard weight-loss programmebo
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
pg/ml | 92.05 (69.45) | 88.25 (37.00)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.8591, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p = 0.0404, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p = 0.0474, Paired t-test

24. Secondary Outcome: 8-HETE at 6 Months
Description: Level of 8-HETE at 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
pg/ml | 70.10 (28.45) | 82.88 (36.02)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.3187, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p = 0.0482, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p = 0.0394, Paired t-test

25. Secondary Outcome: 5-HETE at 2 Months
Description: Level of 5-HETE at 2 months
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
pg/ml | 512.39 (362.39) | 399.09 (126.57)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.2813, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p = 0.4421, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p = 0.3198, Paired t-test

26. Secondary Outcome: 5-HETE at 6 Months
Description: Level of 5-HETE at 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
pg/ml | 313.75 (104.23) | 369.10 (149.68)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.2792, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p = 0.1034, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p = 0.9898, Paired t-test

27. Secondary Outcome: TXB2 at 2 Months
Description: Level of TXB2 at 2 months
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
pg/ml | 177.96 (249.02) | 149.31 (123.06)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.7047, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p = 0.4749, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p = 0.6014, Paired t-test

28. Secondary Outcome: TXB2 at 6 Months
Description: Level of TXB2 at 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
pg/ml | 132.57 (76.49) | 148.01 (71.79)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.5932, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p = 0.7140, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p = 0.5827, Paired t-test

29. Secondary Outcome: PGE2 at 2 Months
Description: Level of PGE2 at 2 months
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
pg/ml | 16.58 (36.39) | 5.58 (10.77)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.2894, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p = 0.2128, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p = 0.0823, Paired t-test

30. Secondary Outcome: PGE2 at 6 Months
Description: Level of PGE2 at 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
pg/ml | 28.73 (57.82) | 13.31 (15.46)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.3450, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p = 0.1365, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p = 0.0073, Paired t-test

31. Secondary Outcome: LTB4 at 2 Months
Description: Level of LTB4 at 2 months
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
pg/ml | 43.41 (128.46) | 1.49 (5.58)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.2333, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p = 0.4292, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p = 0.3356, Paired t-test

32. Secondary Outcome: LTB4 at 6 Months
Description: Level of LTB4 at 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
pg/ml | 13.34 (18.30) | 16.31 (18.99)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.6830, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p = 0.8625, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p = 0.0068, Paired t-test

33. Secondary Outcome: 17-HDOHE at 2 Months
Description: Level of 17-HDOHE at 2 months
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
pg/ml | 172.24 (123.32) | 213.17 (109.31)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.3694, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p = 0.0291, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p = 0.0402, Paired t-test

34. Secondary Outcome: 17-HDOHE at 6 Months
Description: Level of 17-HDOHE at 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
pg/ml | 177.95 (120.73) | 286.03 (214.13)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.1226, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p = 0.0472, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p = 0.0197, Paired t-test

35. Secondary Outcome: 14-HDOHE at 2 Months
Description: Level of 14-HDOHE at 2 months
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
pg/ml | 3320.96 (2520.22) | 3423.64 (1452.23)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.8969, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p = 0.7218, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p = 0.4536, Paired t-test

36. Secondary Outcome: 14-HDOHE at 6 Months
Description: Level of 14-HDOHE at 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
pg/ml | 2760.07 (3984.42) | 2575.02 (1833.92)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.8765, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p = 0.5114, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p = 0.0237, Paired t-test

37. Secondary Outcome: 7-HDOHE at 2 Months
Description: Level of 7-HDOHE at 2 months
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
pg/ml | 118.46 (42.42) | 140.10 (59.71)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.2914, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p = 0.5594, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p = 0.2532, Paired t-test

38. Secondary Outcome: 7-HDOHE at 6 Months
Description: Level of 7-HDOHE at 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
pg/ml | 149.72 (47.26) | 190.58 (56.36)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.0528, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p = 0.1920, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p = 0.0011, Paired t-test

39. Secondary Outcome: 4-HDOHE at 2 Months
Description: Level of 4-HDOHE at 2 months
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
pg/ml | 298.81 (102.32) | 346.78 (130.19)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.2999, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p = 0.5184, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p = 0.0564, Paired t-test

40. Secondary Outcome: 4-HDOHE at 6 Months
Description: Level of 4-HDOHE at 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
pg/ml | 207.26 (94.35) | 306.24 (171.67)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.0783, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p = 0.1263, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p = 0.6484, Paired t-test

41. Secondary Outcome: RVD2 at 2 Months
Description: Level of RVD2 at 2 motnhs
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
pg/ml | 29.15 (37.23) | 23.16 (39.62)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.6896, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p = 0.0980, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p = 0.3526, Paired t-test

42. Secondary Outcome: RVD2 at 6 Months
Description: Level of RVD2 at 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
pg/ml | 31.08 (33.48) | 31.73 (44.41)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.9662, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p = 0.1450, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Test type: Superiority or Other; p = 0.3811, Paired t-test

43. Secondary Outcome: PD1 at 2 Months
Description: Level of PD1 at 2 months
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
pg/ml | 3.70 (4.99) | 6.06 (5.69)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.2643, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p = 0.0761, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p = 0.1342, Paired t-test

44. Secondary Outcome: PD1 at 6 Months
Description: Level of PD1 at 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
pg/ml | 4.51 (3.11) | 6.31 (3.03)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.1410, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p = 0.3774, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Test type: Superiority or Other; p = 0.1811, Paired t-test

45. Secondary Outcome: 7SMAR1 at 2 Months
Description: Level of 7SMAR1 at 2 months
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
pg/ml | NA (NA) — 7SMAR1 at 2 months was below limits of detection | NA (NA) — 7SMAR1 at 2 months was below limits of detection
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p < 0.0001, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p < 0.0001, Paired t-test

46. Secondary Outcome: 7SMAR1 at 6 Months
Description: Level of 7SMAR1 at 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
pg/ml | 5.52 (8.81) | 7.35 (8.52)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.5893, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p = 0.0431, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p = 0.0066, Paired t-test

47. Secondary Outcome: 7RMAR1 at 2 Months
Description: Level of 7RMAR1 at 2 months
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
pg/ml | NA (NA) — 7RMAR1 at 2 months was below limits of detection | NA (NA) — 7RMAR1 at 2 months was below limits of detection
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p < 0.0001, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p < 0.0001, Paired t-test

48. Secondary Outcome: 7RMAR1 at 6 Months
Description: Level of 7RMAR1 at 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
pg/ml | 6.01 (3.29) | 6.05 (6.95)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.9850, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 6 month data; Test type: Superiority or Other; p = 0.0049, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Test type: Superiority or Other; p = 0.0062, Paired t-test

49. Secondary Outcome: Sum of Proinflammatory Mediators at 2 Months
Description: sum of proinflammatory mediators at 2 months
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
pg/ml | 7470.14 (4105.76) | 5842.09 (1944.08)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.1946, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p = 0.2337, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p = 0.9188, Paired t-test

50. Secondary Outcome: Sum of Proresolving Mediators at 2 Months
Description: sum of proresolving mediators at 2 months
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
pg/ml | 3943.32 (2545.83) | 4152.90 (1545.52)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.7964, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p = 0.7680, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p = 0.5669, Paired t-test

51. Secondary Outcome: Proresolution Index
Description: Proresolution index is the ratio of sum of proresolving mediators/sum of proinflammatory mediators
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 15 | 14
ratio | 0.55 (0.20) | 0.72 (0.19)
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.0320, ANCOVA
Statistical Analysis 2: Comparison: Control; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p = 0.0220, Paired t-test
Statistical Analysis 3: Comparison: Omega-3 DHA; Within-group comparisons between the baseline and 2 month data; Test type: Superiority or Other; p = 0.4563, Paired t-test

52. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: Number of Participants with Adverse Events as a Measure of Safety and Tolerability of standardized weight-loss programme (PronoKal® Method)and Safety and Tolerability of DHA Supplements
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Control | Omega-3 DHA
Number analyzed (Participants) | 17 | 17
participants
  Blood and lymphatic system disorders (hypotension) | 2 | 0
  Gastrointestinal disorders | 7 | 7
  General disorders | 2 | 6
  Musculoskeletal and connective tissue disorders | 2 | 1
  Nervous system disorders (migraine, cephalea) | 0 | 2
  Skin and subcutaneous tissue disorders (hair loss) | 1 | 3
Statistical Analysis 1: Comparison: Control vs Omega-3 DHA; Between-Group Comparison; Test type: Superiority or Other; p = 0.72828, Fisher Exact

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Control | Omega-3 DHA
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 9/17 | 11/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=17) | Omega-3 DHA (N=17)
Gastrointestinal Disorders (Gastrointestinal disorders) | 7 (7) | 7 (9) — Constipation, vomiting, diarrhea, stomachache, heartburn
Musculokeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) — Muscle pain, bone pain, muscular weakness
General Disorders (General disorders) | 2 (2) | 6 (13) — Halitosis, asthenia, heaviness, tiredness, cramps, hyperuricemia
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 2 (2) | 0 (0) — Hypotension
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) — Hair loss, urticaria
Nervous System disorders (Nervous system disorders) | 0 (0) | 2 (3) — Cephalea, migraine, headache effort

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes